CLINICAL TRIAL: NCT02862847
Title: Study of the Prevalence of Cosavirus and Salivirus Infections, Two New Genera of Picornaviridae, In Infants
Acronym: COSALE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DE ROUGEMONT AOI 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Gastro entérite

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- gastroenteritis
  Interventions: Other: stool samples
- control
  Interventions: Other: stool samples

INTERVENTIONS:
Other: stool samples

SUMMARY:
Cosavirus and Salivirus are two new genera of Picornaviridae and are responsible for acute diarrhoea. They have been identified in the pathological stools of infants and immuno-compromised subjects on every continent with prevalences ranging from 2.8% to 8.8% depending on the virus, the cohort and the country studied.

To date, no study on these two viruses has been conducted in France to evaluate the circulation and the pathogenicity of these viruses in subjects with diarrhoea.

The aim of this study is thus to:

* show that these viruses are in circulation in France in infants younger than 5 years old and that the proportions are similar to those reported in the literature.
* confirm the relationship between the diarrhoea and the infection with these viruses.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 5 years
* Children hospitalized or consulting at Dijon CHU during the 12 months of the study for acute gastroenteritis. Acute gastroenteritis is defined by at least 3 soft or liquid stools or at least 3 bouts of vomiting within 24 hours or signs (diarrhoea or vomiting) accompanied by at least 2 additional symptoms among diarrhoea or vomiting, abdominal pain, fever

for controls

* Children younger than 5 years old
* Children hospitalized or consulting at Dijon CHU during the 12 months of the study for any illness without diarrhoea (other than exclusion criteria).

Exclusion Criteria:

* Persons without national health insurance cover
* Children older than 5 years.
* Children presenting chronic diarrhoea (> 2 weeks) (e.g. Crohn and UC)
* Children with immune deficiency.
* Children with nosocomial gastroenteritis; the nosocomial aspect will be defined as the onset of acute diarrhoea occurring after the 48th hour after admission

for controls

* Persons without national health insurance cover
* Children older than 5 years.
* Children with chronic diarrhoea (> 2 weeks) (e.g. Crohn and UC)
* Children with immune deficiency.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children de moins de 5ans présentant ou non un épisode de gasto entérite
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of viruses detected | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France